CLINICAL TRIAL: NCT04014387
Title: Treatment of Disturbed Sleep in Progressive Supranuclear Palsy (PSP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20181608
Record Dates: First submitted 2019-04-11; First posted 2019-07-10 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Treatment
MeSH Terms: interventions — suvorexant; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Zolpidem Arm (Active Comparator): Participants will be given one week of Zolpidem.
  Interventions: Drug: Zolpidem
- Suvorexant Arm (Active Comparator): Participants will be given one week of Suvorexant.
  Interventions: Drug: Suvorexant
- Placebo Arm (Placebo Comparator): Participants will be given one week of a placebo pill.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Suvorexant — Suvorexant (Belsomra) is an FDA approved, dual orexin receptor antagonist. It is prescribed for insomnia, reducing time to sleep onset, and to maintain nighttime sleep.
  Other Names: Belsomra
  Arms: Suvorexant Arm
Drug: Zolpidem — Zolpidem (Ambien) is an FDA approved, Benzodiazepine Receptor agonist that has been extensively studied for the treatment of insomnia in older adults. It acts as a sedative and is typically prescribed to treat insomnia, reducing time to sleep onset, but may not alter the ability to maintain sleep.
  Other Names: Ambien
  Arms: Zolpidem Arm
Drug: Placebo oral capsule — Placebo (microcrystalline cellulose) capsules will be used.
  Arms: Placebo Arm

SUMMARY:
Prior research has identified profound sleep disruption in individuals with PSP. Not only were these individuals sleeping relatively short periods at night, they were also not recuperating lost sleep during the day. Research also showed the relative preservation of a series of nuclei key in regulating wake and arousal. Investigators believe that therapeutically targeting wake promoting centers with a specific medication will improve sleep quality and overall well-being in PSP. To study this, investigators will be doing a double blind, within subject, remote clinical trial with 3 conditions: suvorexant- which targets a wake promoting system, zolpidem- a standard hypnotic that engages sleep promoting systems, versus placebo. Each condition will last 1 week and will be separated by a 1 week washout period on no sleep medications. Investigators will measure sleep patterns and daytime symptoms to determine if suvorexant, zolpidem, or both medications are safe and effective for treating sleep disturbances and improving overall well-being in PSP.

ELIGIBILITY:
Inclusion Criteria:

Male or female ≥18 years of age at baseline.

Documentation of a Progressive Supranuclear Palsy diagnosis as evidenced by one or more clinical features consistent with the Progressive Supranuclear Palsy phenotype as described in the Movement Disorder Society criteria or the NINDS-SPSP criteria.

Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Have a diagnosis of PSP verified through co-enrollment in ARTFL, LEFFTDS or 4RTNI, or can show evidence of an accurate diagnosis of PSP to the satisfaction of the study team doctor (e.g. through review of medical records, and/or specific communication with a known medical doctor).

Have an active caregiver who is willing and able to participate in this study

Have a mailing address

Have access to a phone

Have stable medications (aside from sleep-modifying medications) for 4 weeks prior to actively starting the study

Be free of sleep modifying medications for 1 week prior to actively starting the study

Be willing to maintain a stable sleeping environment and their typical daily schedule for the duration of the 6-week study

Resides in a US territory or state covered by our research study team.

Exclusion Criteria:

Are pregnant, breastfeeding, or unwilling to practice birth control if appropriate during participation in the study.

Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Presence of a major psychiatric disorder aside from anxiety or depression.

Presence of a medical condition other than PSP that could account for cognitive deficits (e.g. active seizure disorder, stroke, vascular dementia).

Presence of current substance abuse or substance dependence.

Presence of a significant systemic medical illness (e.g. significant cardiovascular, hematologic, renal, or hepatic disease).

Presence of current medication likely to affect sleep outcomes: benzodiazepine receptor agonists (e.g. Zolpidem), Suvorexant, sedating antipsychotics (e.g. Quetiapine), sedating antihistamines (e.g. Benadryl), low dose sedating antidepressants (e.g. Trazodone, Doxepin), over the counter sleep-inducing medications (e.g. Tylenol-PM), neuroleptics in the phenothiazine and haloperidol families) which 1) the potential participant is not able/willing to stop taking for 1- week prior and for the 6-week duration of the study and/or 2) if removed could have a persistent effect beyond the 1-week wash-out period.

Presence of insulin-dependent diabetes.

History of mental retardation.

Unable to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-02 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency | average each of the 7 nights of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1).
  Change in sleep efficiency (as measured by actigraphy), this is a percentage of the time spent asleep compared to the total time in bed. The range of scores is 0-100, with higher scores associated with better sleep efficiency.
Clinical Global Impression | 7th day of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1).
  Change in Clinical Global Impression (CGI-C), this is a series of questions for the participant and caregiver which the neurologist utilizes to give a score of disease affects across a series of domains, which produces a single change score referenced to the baseline Clinical Global Impression of Disease Severity (CGI-ds). The range of scores is 1-7, with lower scores associated with better health.

SECONDARY OUTCOMES:
Medication Satisfaction | 7th day of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6)
  Differences in satisfaction with the medication being taken. The Medication Satisfaction Scale is a study-specific customized satisfaction questionnaire of 3 questions each with a 5-point likert scale. The total range of scores is 3-15, with higher scores associated with greater medication satisfaction.
Adverse Events | total of events across the 7 days/nights of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1).
  The difference in the number of adverse events across each assessment week. The range of scores is 0 - undetermined, with greater scores associated with greater adverse events.
Alertness | 7th day of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1)
  Change in alertness, which is assessed using question 8 of the Mayo Sleep Questionnaire - Informant. The range of scores is 0-10 with higher scores associated with greater alertness.
Sleepiness | 7th day of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1).
  Change in sleepiness, which is assessed using the Epworth Sleepiness Scale. The range of scores is 0-24 with higher scores associated with increased sleepiness.
Insomnia | 7th day of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1).
  Change in subjectively reported insomnia assessed using the Insomnia Severity Index. The range of scores is 0-28 with higher scores associated with increased levels of insomnia.
Anxiety | 7th day of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1).
  Change in anxiety levels assessed using the Generalized Anxiety Disorder - 7 (GAD-7) scale. The range of scores is 0-21 with higher scores associated with greater anxiety.
Depression | 7th day of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1).
  Change in depression assessed using the PHQ-9 scale. The range of scores is 0-27 with higher scores associated with greater depression.
Quality of Life Survey | 7th day of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1).
  Change in quality of life using the PSP Quality of life survey (PSP-QoL) , which assesses subjective quality of life specifically in individuals with Progressive Supranuclear Palsy. The range of scores is 0-100 with higher scores associated with poorer quality of life.
Functionality | 7th day of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1).
  Change in functionality is assessed using the Tau functional scale. This is a questionnaire, which both the patient and caregiver work together to complete. The total range of scores is 0-124 with subscores for "motor experiences of daily living" (0-48 points), "Language/cognitive/behavioral" concerns (0-52) and "Other non-motor experiences of daily living" (0-24). In all cases, greater scores are associated with decreased independent functionality in those domains.
Cognition | 7th day of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1)
  Change in cognition will be assessed using working memory measures of digits forward and digits backward, and executive function measures of categorical fluency and verbal fluency. The range of scores for digits forward and digits backward is 0-16 each, with higher scores indicating better cognition. The likely range of scores for the fluency measures are 0-60 with higher scores associated with better executive function. Rule violations and repetitions are also counted and scored with greater scores in these domains associated with poorer cognition.
Slow wave sleep | average of 5th-7th night of treatment for each of the two hypnotic drugs and placebo (weeks 2, 4 and 6) compared to baseline (week 1).
  Change in slow wave sleep will be assessed using a mobile EEG monitor called the Sleep Profiler (Advanced Brain Monitoring, Inc.). The amount of slow wave sleep will be measured as a percent of total sleep time, so the range of scores will be 0-100, with higher scores associated with greater amounts of slow wave sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Neylan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California- San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walsh CM, Ruoff L, Walker K, Emery A, Varbel J, Karageorgiou E, Luong PN, Mance I, Heuer HW, Boxer AL, Grinberg LT, Kramer JH, Miller BL, Neylan TC. Sleepless Night and Day, the Plight of Progressive Supranuclear Palsy. Sleep. 2017 Nov 1;40(11):zsx154. doi: 10.1093/sleep/zsx154. PMID 29029214